CLINICAL TRIAL: NCT01471691
Title: Phase I/II, Open-label, Study of Intravitreal RAnibizumab 0.5MG, or High Dose 1.0mg for Retinal Vein Occlusions With rEfractory Macular Edema Previously Receiving iNtravitreal Bevacizumab (RAVEN)
Brief Title: Intravitreal Ranibizumab 0.5MG, or 1.0mg for RVO With Macular Edema Previously Receiving Bevacizumab
Acronym: RAVEN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanscom, Thomas, M.D. (Individual)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML27847
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Branch Retinal Vein Occlusion; Central Retinal Vein Occlusion; Macular Edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravitreal ranibizumab 0.5mg (Experimental)
  Interventions: Drug: ranibizumab 0.5mg
- intravitreal ranibizumab 1.0mg (Experimental)
  Interventions: Drug: ranibizumab 1.0mg

INTERVENTIONS:
Drug: ranibizumab 0.5mg — Standard dose
  Other Names: Lucentis
  Arms: intravitreal ranibizumab 0.5mg
Drug: ranibizumab 1.0mg — High dose
  Other Names: Lucentis
  Arms: intravitreal ranibizumab 1.0mg

SUMMARY:
This study examines two doses of Ranibizumab (0.5mg and 1.0mg) for the treatment of macular edema secondary to retinal vein occlusion in patients that have previously failed treatment with other macular edema treatments including bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* CRVO or BRVO diagnosis
* For CRVO, clinical evidence of perfused central retinal vein occlusion. A CRVO is defined as an eye that has retinal hemorrhages and a dilated retinal venous system in all 4 quadrants. Other evidence of a CRVO may include telangiectatic capillary bed and collateral vessels at the optic nerve head.
* Central macular edema present on clinical examination and OCT testing with a central point thickness and/or central 1mm subfield thickness > 300 microns after at least 3 months of bevacizumab or steroid therapy.
* Visual acuity score greater than or equal to 19 letters (20/400) and less than or equal to 73 letters (20/40) by the ETDRS visual acuity protocol.
* Patients must demonstrate that they are no longer improving on bevacizumab or intravitreal steroid therapy (i.e. no improvement in acuity in 2 consecutive visits)
* BRVO patients treated with grid laser must show residual edema three months following latest laser treatment
* Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or known to be pregnant; also pre-menopausal women not using adequate contraception.
* Participation in another ocular investigation or trial simultaneously
* Any condition that, in the opinion of the investigator, would preclude participation in the study (e.g. chronic alcoholism, drug abuse)
* Significant diabetic retinopathy (greater than moderate NPDR) or macular edema associated with diabetic retinopathy
* An eye that, in the investigator's opinion, has no chance of improving in visual acuity following resolution of macular edema (e.g. presence of subretinal fibrosis or geographic atrophy or severe epiretinal membrane)
* Presence of another ocular condition that may affect the visual acuity or macular edema during the course of the study (e.g. AMD, uveitis, Irvine-Gas)
* Evidence of neovascularization of the iris or retina (presence of ischemic CRVO/BRVO)
* Evidence of central atrophy or fibrosis in the study eye
* Presence of substantial cataract, one that might decrease the vision by 3 or more lines of vision at sometime during the study.
* History of grid/focal laser or panretinal laser in the study eye in the previous three months
* History of vitreous surgery in the study eye
* History of use of intravitreal, peribulbar, or retrobulbar steroids within three months of the study.
* History of cataract surgery within 6 months of enrollment.
* History of YAG capsulotomy within 2 months of the surgery.
* Visual acuity <20/400 in the fellow eye
* Uncontrolled glaucoma (pressure >30) despite treatment with glaucoma medications.
* History of cerebral vascular accident or myocardial infarction within 3 months prior to Day 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O'Hearn, MD, Principal Investigator — Thomas Hanscom AMC
Locations (4):
- United States (4):
  - South Coast Retina, Huntington Beach, California
  - South Coast Retina, Long Beach, California
  - Thomas Hanscom AMC, Santa Monica, California
  - South Coast Retina, Torrance, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravitreal Ranibizumab 0.5mg: ranibizumab 0.5mg: Standard dose Patients were given six months of monthly treatment with the standard 0.5mg ranibizumab dose, followed by six months of evaluation and PRN treatment based upon pre-specified criteria.
- Intravitreal Ranibizumab 1.0mg: ranibizumab 1.0mg: High dose Patients were given six months of monthly treatment with the 1.0mg ranibizumab dose, followed by six months of evaluation and PRN treatment based upon pre-specified criteria.
Period: Overall Study
Arm/Group | Intravitreal Ranibizumab 0.5mg | Intravitreal Ranibizumab 1.0mg
Started | 8 | 6
Completed | 8 | 5
Not Completed | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravitreal Ranibizumab 0.5mg | Intravitreal Ranibizumab 1.0mg | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (5.0) | 78 (5.0) | 75 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline BCVA
Description: Vision was measured using a standard ETDRS chart at baseline and each subsequent monthly visit.
Time Frame: Baseline to month 6
Measure: Mean (Standard Deviation); unit: Letters (ETDRS chart)
Arm/Group | Intravitreal Ranibizumab 0.5mg | Intravitreal Ranibizumab 1.0mg
Number analyzed (Participants) | 8 | 5
Letters (ETDRS chart) | 14 (10) | 5 (6)

2. Secondary Outcome: Mean Change From Baseline in Center Point Thickness
Time Frame: months 1-12
Reporting Status: Not Posted

3. Secondary Outcome: Change in Mean Best Corrected Visual Acuity From Baseline
Time Frame: months 1-12
Reporting Status: Not Posted

4. Secondary Outcome: Percentage of Patients With CFT Less Than 300um
Time Frame: Month 6 and 12
Reporting Status: Not Posted

5. Secondary Outcome: Excess Foveal Thickness
Time Frame: Month 6 and 12
Reporting Status: Not Posted

6. Secondary Outcome: Total Number of Ranibizumab Injections
Time Frame: month 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intravitreal Ranibizumab 0.5mg | Intravitreal Ranibizumab 1.0mg
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal Ranibizumab 0.5mg (N=8) | Intravitreal Ranibizumab 1.0mg (N=6)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Patient developed breast cancer during trial. It was treated by her oncologist. Not felt to be secondary to Ranibizumab.
Ruptured Retinal Macroaneurysm (Ear and labyrinth disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes